CLINICAL TRIAL: NCT01075542
Title: Efficacy and Cost-effectiveness of Toric Intraocular Lenses in Correcting Astigmatism in Cataract Surgery: a Randomised Clinical Trial
Brief Title: Astigmatism Management in Cataract Surgery With the AcrySof Toric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 082099
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Astigmatism
Keywords: Corneal astigmatism; Intraocular lens
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toric intraocular lens (Experimental): Bilateral Toric intraocular lens implantation in cataract surgery
  Interventions: Device: AcrySof Toric intraocular lens, model SN60TT
- Monofocal intraocular lens (Other): Bilateral Monofocal intraocular lens implantation in cataract surgery
  Interventions: Device: AcrySof Monofocal IOL, model SN60AT

INTERVENTIONS:
Device: AcrySof Toric intraocular lens, model SN60TT — The lens is made of foldable acrylic material and is implanted in the capsular bag
  Arms: Toric intraocular lens
Device: AcrySof Monofocal IOL, model SN60AT — The lens is made of foldable acrylic material and is implanted in the capsular bag
  Arms: Monofocal intraocular lens

SUMMARY:
The purpose of this study is to determine if Toric intraocular lens implantation in cataract surgery is a more efficient and cost-effective treatment of astigmatism than Monofocal intraocular lens implantation.

DETAILED DESCRIPTION:
A recent innovation in cataract surgery consists of the introduction of toric intraocular lenses (IOLs) that can correct corneal astigmatism. It offers the opportunity for patients with substantial astigmatism to achieve optimal distance vision without using spectacles. Good near vision may subsequently be achieved with low-cost reading glasses. The current practice of non-toric IOL implantation in astigmatic patients warrants the use of expensive bifocal or multifocal spectacles with cylinder correction to achieve good distance and near vision.

Objective: The primary objective of this study is to compare spectacle independence for distance vision following toric IOL implantation and monofocal intraocular lens (IOL) implantation. The secondary objectives are to compare uncorrected distance vision, residual refractive astigmatism, quality of vision, wavefront aberrations, contrast sensitivity, complication profile, costs of postoperative spectacles and cost-effectiveness.

Study design: Multi-centre randomised clinical trial. Study population: 160 patients with regular corneal astigmatism of at least 1.25 diopters in both eyes who require bilateral cataract surgery.

Intervention: Cataract surgery with implantation of a toric IOL (AcrySof model SN60TT) or an monofocal IOL (AcrySof model SN60AT).

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract
* Bilateral corneal astigmatism (at least 1.25D)
* Predicted residual astigmatism less than 0.5D

Exclusion Criteria:

* Irregular corneal astigmatism or keratoconus
* Fuchs endothelial dystrophy (stage 2)
* Expected postoperative best-corrected visual acuity worse than logMAR +0.3

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Spectacle independency | preop, 3 months and 6 months postop
  Spectacle independency for distance vision

SECONDARY OUTCOMES:
Visual acuity | preop, 1 day, 1 month, 3 months and 6 months postop
Refractive astigmatism | preop, 3 months and 6 months postop
Higher-order wavefront aberrations | preop, 3 months and 6 months postop
Contrast sensitivity | preop, 3 months and 6 months postop
Costs related to intervention | preop, 3 and 6 months postop
  Total cost-analysis, including out-of-hospital costs for patient
Quality of vision | preop, 3 months, 6 months
  Refractive-error related quality of vision

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (3):
- Netherlands (3):
  - Atrium Medical Center, Heerlen, Brunssum, Kerkrade
  - Maastricht University Medical Center, Maastricht
  - Rotterdam Eye Hospital, Rotterdam

REFERENCES:
- [Background] Bauer NJ, de Vries NE, Webers CA, Hendrikse F, Nuijts RM. Astigmatism management in cataract surgery with the AcrySof toric intraocular lens. J Cataract Refract Surg. 2008 Sep;34(9):1483-8. doi: 10.1016/j.jcrs.2008.05.031. PMID 18721707
- [Derived] Visser N, Beckers HJ, Bauer NJ, Gast ST, Zijlmans BL, Berenschot TT, Webers CA, Nuijts RM. Toric vs aspherical control intraocular lenses in patients with cataract and corneal astigmatism: a randomized clinical trial. JAMA Ophthalmol. 2014 Dec;132(12):1462-8. doi: 10.1001/jamaophthalmol.2014.3602. PMID 25256624